CLINICAL TRIAL: NCT00132977
Title: Resynchronization Therapy in Normal QRS (RethinQ) Clinical Investigation
Brief Title: RethinQ Study - Evaluating Pacing in Heart Failure Patients
Acronym: RethinQ
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G050084
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
Keywords: Cardiac Resynchronization Therapy; Heart Failure; Mechanical Dyssynchrony
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy

SUMMARY:
Patients with heart failure have a pumping action of the ventricles in which one ventricle contracts before the other ventricle. This uncoordinated (unsynchronized) pumping is due to a delay in the stimulation of the left ventricle because of its increased size. Pacing both the right and the left side of the heart (or cardiac resynchronization therapy [CRT]) has been proven to be effective in the treatment of heart failure (HF). Current market-approved devices combine both pacing (CRT) and shocking (implantable cardioverter defibrillator [ICD]) therapy for patients who have severe heart failure and are at risk for developing life-threatening heart rhythms. These devices provide an electrical pacing stimulus to both ventricles and may help the heart contract in a more coordinated way and improve heart failure symptoms.

The investigational portion of this trial involves the implantation of a market-approved CRT implantable cardioverter defibrillator (CRT-D) system in patients who do not meet the current criteria for a CRT implant. In order to receive a CRT-D implant today, patients must have heart failure symptoms, have a weakened heart muscle, and have uncoordinated pumping of the heart. To demonstrate this uncoordinated pumping of the heart, a test (electrocardiogram [ECG]) is done. It is believed that by using a different test (echocardiogram) to measure whether this uncoordinated pumping is present, more patients will be identified that will benefit from CRT-D therapy. This study will look at whether patients identified by using this echocardiogram test show a benefit from having this CRT-D therapy.

DETAILED DESCRIPTION:
1.0 Problem of Interest

Patients with heart failure have a pumping action of the ventricles in which one ventricle contracts before the other ventricle. This uncoordinated (unsynchronized) pumping is due to a delay in the stimulation of the left ventricle because of its increased size. Pacing both the right and the left side of the heart (or cardiac resynchronization therapy [CRT]) has been proven to be effective in the treatment of heart failure. Current market-approved devices combine both pacing (CRT) and shocking (ICD) therapy for patients who have severe heart failure and are at risk for developing life-threatening heart rhythms. These devices provide an electrical pacing stimulus to both ventricles at the same time and may help the heart contract in a more coordinated way and improve heart failure symptoms.

The investigational portion of this trial involves the implantation of a market-approved CRT implantable cardioverter defibrillator (CRT-D) system in patients who do not meet the current criteria for a CRT implant. In order to receive a CRT-D implant today, patients must have heart failure symptoms, have a weakened heart muscle, and have uncoordinated pumping of the heart. To demonstrate this uncoordinated pumping of the heart, a test (ECG) is done. It is believed that by using a different test (echocardiogram) to measure whether this uncoordinated pumping is present, more patients will be identified that will benefit from CRT-D therapy.

2.0 Study Summary

Testing will be performed to determine if patients are eligible for this study. An EKG (electrical tracing of the heart) will be performed. They will be asked to complete a 6- minute hall walk test that will provide information regarding their ability to exercise and conduct daily activities. An echocardiogram with tissue Doppler imaging (ultrasound of the heart) will be performed to determine how the heart muscle contracts. Results of this echocardiogram will determine if patients are eligible to participate in this study.

The device system that will be implanted consists of a St. Jude Medical CRT-D and three pacing leads (insulted wires that carry electrical energy from the device to the heart). One lead is placed in the upper right chamber of the heart (atrium), a second lead is placed in the lower right chamber of the heart (right ventricle) and the third lead is placed within a vein that runs along the outside of the heart and is positioned at a location near the left lower chamber of the heart (left ventricle).

A randomization visit will occur approximately 14 days after implant. Patients will be randomized (like a flip of a coin) to one of two groups. Each patient will have an equal chance of being randomized to either of the two groups. One group will receive cardiac resynchronization treatment (CRT ON) and the other group will not receive cardiac resynchronization treatment (CRT OFF). Patients in the CRT OFF group can receive cardiac resynchronization treatment at 6 months after randomization if the doctor determines that it is appropriate.

Prior to randomization and programming of the device, the following tests will be completed:

* Quality of Life Questionnaire - contains 21 questions that provide information as to how heart failure affects the patient's daily life.
* EKG
* 6-Minute Hall.
* Cardiopulmonary Exercise Stress Testing (CPX) - measures the amount of oxygen used by your body while exercising on a treadmill and breathing through a special breathing tube
* Echocardiogram

Follow-up visits will occur at 3 and 6 months following randomization and every 6 months thereafter until the end of the study. The tests performed at the randomization visit (Quality of Life Questionnaire, EKG, 6 minute hall walk, CPX and echocardiogram) will be repeated at the 6-month follow-up visit. Additionally, each visit will include a review of the patient's condition and current medications and an evaluation of the CRT-D device.

3.0 How Will the Research Advance Scientific Knowledge and/or Human Health?

It is hoped that by pacing both lower chambers of the heart in these patients that they will feel better. They may be able to do more activities with fewer symptoms. In addition, the information gathered in this study will add to the understanding of treatment options for patients with heart failure.

4.0 What is the Current Standard of Care?

Alternative treatments to the St. Jude Medical CRT-D system (includes the left heart lead) currently available include implantation of a standard ICD system and/or treatment with medications.

ELIGIBILITY:
Inclusion Criteria:

* Have an approved indication for implantation of an ICD.
* Have advanced HF with a New York Heart Association (NYHA) Classification of III, despite receiving optimal pharmacological therapy.
* Have a stable heart failure medical regimen.
* Have a left ventricular ejection fraction (LVEF) <= 35%.
* Have evidence of mechanical dyssynchrony as measured by echocardiography using tissue Doppler imaging or M-mode.
* Have a QRS duration < 130 ms (present in all ECG leads).
* Have the ability to complete exercise stress testing and 6-minute hall walk test, with the only limiting factors being related to cardiac fitness.
* Have the ability to independently comprehend and complete a quality of life questionnaire.
* Have the ability to provide informed consent for study participation and be willing and able to comply with the prescribed follow-up tests and schedule of evaluations.

Exclusion Criteria:

* Have a standard bradycardic indication for pacing.
* Have been previously treated with CRT.
* Have continuous atrial fibrillation [AF] (continuous is defined as AF lasting > 1 month) within 1 year prior to enrollment or have undergone cardioversion for AF in the past month.
* Have the ability to walk > 450 meters during the 6-minute walk test.
* Have a NYHA Classification of I, II or IV.
* Have symptomatic chronic obstructive pulmonary disease (COPD) as it relates to exercise ability.
* Have a classification of Status 1 for cardiac transplantation or consideration for transplantation over the next 6 months.
* Have had a recent myocardial infarction, unstable angina or cardiac revascularization (percutaneous transluminal coronary angioplasty [PTCA] or coronary artery bypass graft [CABG]) within 40 days of enrollment.
* Have had a recent cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 3 months of enrollment.
* Have severe musculoskeletal disorder(s).
* Pregnant or planning for pregnancy in the next 6 months.
* Currently participating in, or have participated in any clinical investigation within the last 30 days (the only exception being that of a registry trial).
* Have a life expectancy of less than 6 months.
* Less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2005-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Cardiac resynchronization therapy (CRT) effectiveness will be evaluated in terms of exercise capacity (peak VO2), as measured by cardiopulmonary exercise testing | 6 months
Safety will be evaluated in terms of survival from CRT-D system-related complications. | 6 months

SECONDARY OUTCOMES:
Quality of Life Questionnaire | 6 months
New York Heart Association (NYHA) Classification | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John Beshai, MD, Study Chair — University of Chicago
Locations (34):
- United States (34):
  - University Hospital University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Arrhythmia Consultants, Scottsdale, Arizona
  - Arkansas Cardiology, PA, Little Rock, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Glendale Memorial Hospital and Medical Center, Glendale, California
  - Scripps Green Hospital, La Jolla, California
  - Mercy General Hospital, Sacramento, California
  - St. Francis Hospital and Medical Center, Hartford, Connecticut
  - Shands Jacksonville, Jacksonville, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Unversity of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Iowa Heart Center, Des Moines, Iowa
  - Central Baptist Hospital, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Ingham Regional Medical Center, Lansing, Michigan
  - United Hospital, Saint Paul, Minnesota
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - New York Presbyterian Hospital/Cornell University, New York, New York
  - Mount Sinai Hospital, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Elyria Regional Medical Center, Elyria, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Main Line Health Center/Lankenau Hospital, Wynnewood, Pennsylvania
  - Medical University of Southern California, Charleston, South Carolina
  - Stern Cardiovascular Center, Germantown, Tennessee
  - St. Thomas Hospital, Nashville, Tennessee

REFERENCES:
- [Background] Beshai JF, Grimm R. The resynchronization therapy in narrow QRS study (RethinQ study): methods and protocol design. J Interv Card Electrophysiol. 2007 Sep;19(3):149-55. doi: 10.1007/s10840-007-9156-3. PMID 17899346
- [Result] Beshai JF, Grimm RA, Nagueh SF, Baker JH 2nd, Beau SL, Greenberg SM, Pires LA, Tchou PJ; RethinQ Study Investigators. Cardiac-resynchronization therapy in heart failure with narrow QRS complexes. N Engl J Med. 2007 Dec 13;357(24):2461-71. doi: 10.1056/NEJMoa0706695. Epub 2007 Nov 6. PMID 17986493